CLINICAL TRIAL: NCT05317611
Title: Intravenous Versus Intraperitoneal Instillation of Ondansetron for Decreasing Incidence of Nausea and Vomiting After Laparoscopic Gynecological Surgeries: A Randomized Controlled Study
Brief Title: Intravenous Versus Intraperitoneal Instillation of Ondansetron for Decreasing Incidence of Nausea and Vomiting After Laparoscopic Gynecological Surgeries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Dina Abdelhameed Elsadek Salem, principle investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9286-23-2-2022
Record Dates: First submitted 2022-03-30; First posted 2022-04-08 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Prevention
Keywords: ondansetron; intraperitoneal instillation; laparoscopic gynecological surgeries; postoperative nausea and vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Study the effect of intraperitoneal instillation vs intravenous ondansetron on PONV added to intraperitoneal bupivacaine for enhanced recovery and to decrease incidence of PONV after laparoscopic gynecological surgeries.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessor (anesthesiologist not sharing in the study) will assess outcome parameters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intraperitoneal instillation of ondansetron and bupivacaine (group A) (Active Comparator): Patients will receive intraperitoneal instillation of (100 mg) 40 ml of bupivacaine 0.25 % and (4 mg) 2 ml ondansetron through abdominal ports by simple instillation technique before removal of trocars then clamping of abdominal drains for 1h to avoid drainage of LA.
  Interventions: Drug: Intraperitoneal instillation of ondansetron and bupivacaine
- Intravenous ondansetron and intraperitoneal instillation of bupivacaine (group B) (Active Comparator): Patient will receive intravenous (4 mg) 2 ml ondansetron and intraperitoneal instillation of (100 mg) 40 ml of bupivacaine 0.25 % through abdominal ports by simple instillation technique before removal of trocars then clamping of abdominal drains for 1h to avoid drainage of LA.
  Interventions: Drug: Intravenous ondansetron and intraperitoneal instillation of bupivacaine
- Intraperitoneal instillation of bupivacaine (group C) (Active Comparator): patient will receive intraperitoneal instillation of (100 mg) 40 ml of bupivacaine 0.25 % through abdominal ports by simple instillation technique before removal of trocars then clamping of abdominal drains for 1h to avoid drainage of LA.
  Interventions: Drug: Intraperitoneal instillation of bupivacaine

INTERVENTIONS:
Drug: Intraperitoneal instillation of ondansetron and bupivacaine — The aim is to detect the effect of intraperitoneal instillation of ondansetron for prevention of postoperative nausea and vomiting
  Other Names: Intraperitoneal instillation of zofran and marcaine
  Arms: Intraperitoneal instillation of ondansetron and bupivacaine (group A)
Drug: Intravenous ondansetron and intraperitoneal instillation of bupivacaine — The aim is to detect effect of intravenous ondansetron for prevention of postoperative nausea and vomiting
  Other Names: Intravenous zofran and intraperitoneal instillation of marcaine
  Arms: Intravenous ondansetron and intraperitoneal instillation of bupivacaine (group B)
Drug: Intraperitoneal instillation of bupivacaine — The aim is to detect effect of intraperitoneal instillation of bupivacaine
  Other Names: Intraperitoneal instillation of marcaine
  Arms: Intraperitoneal instillation of bupivacaine (group C)

SUMMARY:
Study the effect of intraperitoneal instillation vs intravenous ondansetron on PONV added to intraperitoneal bupivacaine for enhanced recovery and to decrease incidence of PONV after laparoscopic surgeries.

DETAILED DESCRIPTION:
Laparoscopic surgeries have many advantages e.g., decreasing postoperative pain, better cosmetic, rapid recovery, and better recovery but also, it has side effects e.g., pain, postoperative nausea and vomiting.

There are many risk factors that cause PONV either patient related factors or anesthesia related factors (opioids, inhalational anesthetics, Nitrous oxide and duration of anesthesia) and surgery related factors (intraabdominal, laparoscopic, postoperative pain).

Intraperitoneal instillation of drugs can be used for instillation of LA, opoids, ketamine and antiemetics to provide analgesia and manage side effects of laparoscopic surgery. The mechanism of action of ondansetron is inhibition of presynaptic 5-HT3 receptors that located in the peripheral nervous. Study the effect of intraperitoneal instillation vs intravenous ondansetron on PONV added to intraperitoneal bupivacaine for enhanced recovery and to decrease incidence of PONV after laparoscopic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient.
* Age: 21-60 years old.
* female patients
* Physical status: ASA 1& II.
* BMI = ≤ 35 kg/m2).
* Type of operation: elective laparoscopic gynecological surgeries.

Exclusion Criteria:

* Altered mental state.
* Patients with known history of allergy to the study drugs.
* hepatic, renal impairment or disease , cardiovascular, and respiratory diseases.
* Patients with chronic pain received NSAID or opioid during previous two weeks.
* Patients with history of PONV or motion sickness and patients received antiemetic therapy 24 h before the surgery.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
measure incidence of postoperative nausea and vomiting | 24 hours postoperative
  The number of patient suffering from postoperative nausea and vomiting in each group
measure severity of postoperative nausea and vomiting | 24 hours postoperative
  Simplified Postoperative Nausea and Vomiting Impact Scale (S-PNVIS)
  1. *Frequency of Nausea:*
     * 0: None
     * 1: Occasionally (1-2 times a day)
     * 2: Frequently (3-4 times a day)
     * 3: Constantly (more than 4 times a day)
  2. *Frequency of Vomiting:*
     * 0: None
     * 1: Once a day
     * 2: 2-3 times a day
     * 3: More than 3 times a day
  3. *Impact on Daily Activities:*
     * 0: No impact
     * 1: Mild impact (able to perform most activities)
     * 2: Moderate impact (some activities limited)
     * 3: Severe impact (most activities limited)
       #Scoring
     * *Total Score:* Sum of scores from all 3 items.
     * *Interpretation:* Higher total scores indicate a greater impact of nausea and vomiting on the patient recovery

SECONDARY OUTCOMES:
measure total numbers of rescue antiemetic | all over 24 hours postoperative.
  patients will receive 10 mg intravenous metoclopramide as rescue antiemetic immediately
Duration of hospital stay | 24 hours to 72 hours
  time from PACU discharge till time to discharge home
postoperative pain by Numerical Rating Scale | 0 hour (basal) in PACU, 2, 4, 8, 12, 24 hours postoperative
  10 cm line numbered from 0 to 10, patients instructed to circle the number that represents his/her pain intensity (0=no pain and 10=maximum pain)
total dose of rescue analgesia postoperative | 24 hours postoperative
  total dose of diclofenac as rescue analgesia postoperative
Patient satisfaction | 24 hours postoperative
  degree of satisfaction of the analgesia by using a 5-points Likert-like verbal scale (1 = very dissatisfied analgesia, 2 = dissatisfied analgesia, and 3 = neutral, 4=satisfied analgesia, and 5=very satisfied analgesia)

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of human medicine, Zagazig university hospitals, El Sharkia, Egypt

IPD SHARING:
Plan to Share IPD: No